CLINICAL TRIAL: NCT06163625
Title: The Impact of Working Memory and Reward Markers on DLPFC Activity in Treatment-resistant Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 22-225
Record Dates: First submitted 2023-11-22; First posted 2023-12-11 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-05

CONDITIONS: Major Depressive Disorder; Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant | interventions — Transcranial Magnetic Stimulation; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Depression Group (Experimental)
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation; Behavioral: Research Interview, Questionnaires; Behavioral: Brain Scan; Biological: Saliva Samples
- Control Group (Other)
  Interventions: Behavioral: Research Interview, Questionnaires; Behavioral: Brain Scan; Biological: Saliva Samples

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — For those with depression where medication and psychotherapy have limited benefit, repetitive transcranial magnetic stimulation (rTMS) is an effective treatment. rTMS is a treatment that involves stimulating certain areas of the brain with magnetic field pulses. Over time, the magnetic field pulses can gradually change the activity level of the stimulated brain region. This can be helpful in treating some kinds of psychiatric and neurological disorder, including MDD.
  Arms: Depression Group
Behavioral: Research Interview, Questionnaires — Research Interview: A study team member will meet the participant to ask questions regarding the degree of depression at the beginning of the study. This interview will take approximately 30 minutes.
  Research Questionnaires: A study team member will ask the participant to complete questionnaires assessing the severity of the participant's depression, daily activities, personality/traits, and quality of life. Questionnaires will be completed via pen and paper at each visit. These questionnaires will take approximately 90 minutes to complete.
Behavioral: Brain Scan — The participant will be asked to undergo a magnetic resonance imaging (MRI) scan to look at the structure and function of their brain. The functional MRI measures the level of blood flow to areas of the brain associated with mood and behaviour, and the participant will be asked to complete two behavioural games while they are in the scanner. During the scan, the participant will be required to lie on a table within the cylindrical tube of the MRI scanner in order to complete the scan. This will result in limited movement for the duration of the scan. The scan will take approximately 60 minutes, and there will be a recovery period for 40 minutes. The participant will be given instructions about these tasks outside of the scanner. This brain scan will happen at St. Michael's Hospital.
Biological: Saliva Samples — The participant will be asked to provide six 1mL saliva samples during the MRI scan and recovery period so that the investigators can measure molecular markers associated with depression. In order to provide the sample, the investigators will collect their saliva using a cotton swab and test tube. Each sample should take no more than 5 minutes.

SUMMARY:
Major Depressive Disorder (MDD) is a very common illness that is usually treated with antidepressant medication. Depression can be caused by many things such as childhood experiences, genetics, and changes in the way the body and brain function. For those with depression where medication and psychotherapy have limited benefit, repetitive transcranial magnetic stimulation (rTMS) is an effective treatment. rTMS is a treatment that involves stimulating certain areas of the brain with magnetic field pulses. Over time, the magnetic field pulses can gradually change the activity level of the stimulated brain region. This can be helpful in treating some kinds of psychiatric and neurological disorder, including MDD.

It is not fully known how rTMS changes brain activity to improve symptoms of depression. However, certain brain areas responsible for behaviours impacted by depression are underactive in those with depression. One of those brain regions called the dorsolateral prefrontal cortex (DLPFC), and the investigators will target this region using rTMS. By increasing the activity of these regions, rTMS could potentially improve depression symptoms. For participants receiving rTMS, the investigators will be using the participant's brain scan to better understand brain activity of the brain region stimulated by rTMS before and after treatment.

In this study, the investigators will be collecting detailed information about participants' psychiatric history and depression symptoms, as well as brain scans and saliva samples. The saliva samples will undergo proteomic (having to do with proteins) analyses to identify biological markers ("biomarkers": biological features (e.g.: gene, protein) that can be measured to indicate factors related to rTMS response. The investigators' goal is to use this information to help us understand whether improvement to rTMS depends on brain activity or proteomic factors localized to two specific behaviours impacted by depression: reward processing and working memory (the capacity to hold information temporarily, such as holding a person's address in mind while listening to instructions about how to get there).

ELIGIBILITY:
Inclusion Criteria:

Depressed Participants:

1. Between the ages of 18 and 65 years old.
2. Capable of giving voluntary and informed consent.
3. Fluent in English.
4. Meet Diagnostic and Statistical Manual criteria for single or recurrent Major Depressive Disorder (current major depressive episode), confirmed via the Mini-International Neuropsychiatric Interview (MINI).
5. Moderate to severe depression severity, defined as a 17-item Hamilton Depression Rating Scale260 score ≥ 18.
6. Have failed to achieve a clinical response to an adequate dose of an antidepressant based in an Antidepressant Treatment History Form (ATHF) score ≥ 3 in the current episode, or have been unable to tolerate at least 2 separate trials of antidepressants of inadequate dose and duration (AHTF = 1 or 2)
7. Have had no initiation or dose change in any psychotropic medication in the four weeks prior to screening.
8. If participating in psychotherapy, must have been in stable treatment for at least 3 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions, or the therapeutic focus over the duration of the study.
9. Can adhere to the study schedule.

Nondepressed Participants:

1. Between the ages of 18 and 65 years old.
2. Capable of giving voluntary and informed consent.
3. Fluent in English.
4. No current or previous history of psychiatric diagnoses.
5. Absent/non-clinical depression severity, defined as a 17-item Hamilton Depression Rating Scale260 < 8.
6. No history of antidepressant use, as measured by the ATHF.

Exclusion Criteria:

All Participants:

1. Are pregnant/lactating.
2. Acute suicidality, defined as a score >3 on the 17-item Hamilton Depression Rating Scale, Item #3.
3. A MINI-confirmed diagnosis of bipolar disorder, or another comorbidity (e.g., obsessive-compulsive disorder, post-traumatic stress disorder) that is primary in severity and disability relative to their MDD.
4. Other major medical comorbidities requiring immediate investigation or treatment, cardiac pacemaker, or implanted medication pump.
5. Lifetime history of psychosis, including schizophrenia, schizoaffective disorder, delusional disorder, or current psychotic symptoms.
6. Drug abuse or dependence within the last 6 months, excluding caffeine and nicotine.
7. Contraindication to receiving the rTMS (e.g. history of seizure, cochlear implants, benzodiazepine use (lorazepam or equivalent daily dose >2mg daily), cardiac pacemaker, implanted neurostimulator, significant head trauma with loss of consciousness for greater than or equal to 5 minutes).
8. Electroconvulsive therapy (ECT) within the current depressive episode.
9. Presence of contraindications for MRI, including metallic implants.
10. Have any significant neurological disorder or insult including, but not limited to: any condition likely to be associated with increased intracranial pressure, space occupying brain lesion, any history of seizure except those therapeutically induced by ECT, cerebral aneurysm, Parkinson's disease, Huntington's chorea, multiple sclerosis, dementia, significant head trauma with loss of consciousness for greater than or equal to 5 minutes.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression | Week 0 to End of Treatment (up to 8 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Unity Health Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No